CLINICAL TRIAL: NCT02991807
Title: A Randomized Double-Blind Controlled Trial of Everolimus in Individuals With PTEN Mutations (RAD001XUS257T)
Brief Title: RAD001 and Neurocognition in PTEN Hamartoma Tumor Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Office of Rare Diseases (ORD) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH); Novartis Pharmaceuticals (Industry); PTEN Research (Unknown); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Mustafa Sahin, Director, Translational Neuroscience Center/ Professor of Neurology, Harvard Medical School, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-P00020332; 1U54NS092090 (NIH)
Record Dates: First submitted 2016-12-02; First posted 2016-12-14 (Estimated); Results first posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: PTEN Gene Mutation; PTEN Hamartoma Tumor Syndrome
Keywords: PTEN; PTEN Gene Mutation; PTEN Hamartoma Tumor Syndrome; Autism; Intellectual Disability; Neurocognition; Afinitor; Everolimus; RAD001
MeSH Terms: conditions — Hamartoma Syndrome, Multiple; Autistic Disorder; Intellectual Disability | interventions — Everolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RAD001 (Experimental): RAD001 is formulated as tablets of 5.0 mg or 2.5mg strength, blister-packed under aluminum foil in units of 10 tablets and dosed on a regular basis.
  Interventions: Drug: RAD001
- Placebo (Placebo Comparator): Matching placebo will be provided as a matching tablet and will also be blister packed under aluminum foil in units of 10.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RAD001 — RAD001 is formulated as tablets of 5.0 mg strength, blister-packed under aluminum foil in units of 10 tablets and dosed on a regular basis. RAD001 tablets should be opened only at the time of administration as drug is both hygroscopic and light-sensitive.
  Patients will be instructed to take 4.5 mg/m2 of RAD001 orally with a glass of water at regular intervals at the same time (delete: each day) in the morning after a light, nonfat breakfast.
  Other Names: Everolimus; Afinitor
  Arms: RAD001
Drug: Placebo — Matching placebo will be provided as a matching tablet and will also be blister packed under aluminum foil in units of 10. Matching placebo tablets should be opened only at the time of administration as drug is both hygroscopic and light-sensitive.
  Patients will be instructed to take 4.5 mg/m2 of the matching placebo orally with a glass of water at regular intervals at the same time (delete: each day) in the morning after a light, nonfat breakfast.
  Arms: Placebo

SUMMARY:
Phosphatase and TENsin homolog (PTEN) gene germline mutations are associated with a spectrum of clinical manifestations characterized by neurocognitive deficits, intellectual disability, autism symptomatology, skin lesions, macrocephaly, hamartomatous overgrowth of tissues, and an increased risk of cancers. Investigators are conducting research to evaluate the potential safety and efficacy of RAD001 (everolimus) in this patient population, and the potential neurocognitive benefits from treatment with RAD001 or placebo for a six month period. The investigators hope this trial will lead to a better understanding of PTEN and to new forms of treatment that may benefit children and adults with PTEN in the future.

DETAILED DESCRIPTION:
This is a signal seeking Phase I/II 6-month, randomized, double-blind placebo-controlled trial of everolimus in individuals, ages 5 to 45 years with a PTEN mutation, with safety and neurocognition as the primary endpoints.

Participant's or a legal guardian will need to sign an informed consent prior to enrollment in the study. To determine eligibility participants will undergo a series of screening tests and safety measures. If determined to be eligible for the blinded phase of the study, participants will be randomly assigned to take either the study drug or a placebo (pill with no medicine).

The blinded phase of the study involves about eight visits, five of which will occur at the study site, and three of which will be conducted over the phone. These visits will take place over a six month period. Study visits will vary in length. Baseline, three month and six month visits may last up to 8 hours, if optional measures are done, while all other visits will be less than 2 hours. The study visits include blood draws, general health exams, and neuropsychological assessments. The study will also include optional eye-tracking, EEG and auditory evoked potential (AEP) measures, and the collection of microbiome/mycobiome and biomarker blood sample. There is no fee to participate in this study. The study drug will be provided at no charge during the study.

After the 6 month treatment phase, individuals who were randomly assigned to take placebo will be offered inclusion in a 6 month open label phase where the study drug will be provided at no charge. The open label phase assessments will be similar to those done in the blinded phase, but patients/families will only need to return to the study site three times during this phase.

Participants will receive a developmental assessments report after completing the study. After all study data has been analyzed, patients and families will also be informed of the overall results. Treatment on this study may or may not improve an individual's learning skills (neurocognition) or behavior. We hope that future patients and families will benefit from what is learned by this study.

Specific Aims /Objectives Primary objective

-To evaluate the safety of everolimus compared with placebo in patients with PTEN mutations focusing on NCI CTCAE Grade 3 and 4 adverse events, serious adverse events, and Grade 3 and 4 laboratory toxicities.

Secondary objectives

-To evaluate the efficacy of everolimus on neurocognition and behavior in inividuals with PTEN mutations compared to placebo as measured by standardized, direct and indirect neurocognitive tools and behavioral measures.

ELIGIBILITY:
Double-Blind Inclusion Criteria

1. Male and female outpatients between 5 and 45 years of age (inclusive);
2. Pathogenic PTEN mutation confirmed by clinical genetic testing;
3. Participant must be able to complete one of the following three standardized assessments: Conners' Continuous Performance Tasks (CPT-3-mean reaction time), Stanford Binet (SB-5; working memory), or the Purdue Pegboard Test;
4. Performance below the age-adjusted population mean on at least one of the above standardized measure: attention (CPT-3, mean reaction time), working memory (SB5), or fine motor skills (Purdue Pegboard Test; either dominant hand, non-dominant hand, or both hands);
5. Adequate bone marrow function as shown by:

   1. platelets ≥ 80,000/mm3
   2. absolute neutrophil count ≥ 1,000/mm3
   3. hemoglobin ≥ 9 g/dL
6. Adequate liver function as shown by:

   1. Total serum bilirubin < 1.5 x ULN
   2. AST and ALT levels < 2.5 x ULN
   3. INR ≤ 2
7. Adequate renal function: serum creatinine < 1.5 x ULN,
8. Signed informed consent obtained prior to any screening procedures;
9. Individuals on psychotropic and anti-epileptic medications should maintain a stable dose for at least 2 months prior to the screening visit;
10. Negative serum pregnancy test for females at screening and no plans to become pregnant or conceive a child while participating in the study. The effects of mTOR inhibitors on the developing fetus at the doses used in this study are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for the duration of the study. Estrogen-containing oral contraceptives are not recommended in women enrolled in this study. Abstinence or two effective non-estrogen or barrier methods of contraception (such as condoms + spermicidal foam) must be used;
11. No anticipated changes in the frequency and intensity of existing interventions such as behavioral and developmental treatments, in home services, and speech therapy;
12. No planned changes in school placement;
13. For individuals under 18 or who are otherwise incapable, there must be an available caregiver who can reliably bring subject to clinic visits and provide trustworthy data
14. Able to communicate fluently in English

Double-Blind Exclusion Criteria

1. Patients currently receiving anticancer therapies or who have received anticancer therapies within 4 weeks of the start of Everolimus (including chemotherapy, radiation therapy, antibody based therapy, etc.);
2. Known intolerance or hypersensitivity to Everolimus or other rapamycin analogs (e.g. sirolimus, temsirolimus);
3. Known impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral Everolimus;
4. Uncontrolled diabetes mellitus as defined by HbA1c >8% despite adequate therapy. Patients with a known history of impaired fasting glucose or diabetes mellitus (DM) may be included, however blood glucose and antidiabetic treatment must be monitored closely throughout the trial and adjusted as necessary;
5. Patient with uncontrolled hyperlipidemia: fasting serum cholesterol > 300 mg/dL OR >7.75 mmol/L AND fasting triglycerides > 2.5 x ULN.
6. Patients who have any severe and/or uncontrolled medical or psychiatric conditions (see section 4.6 for additional details)
7. Chronic treatment with corticosteroids or other immunosuppressive agents. Topical or inhaled corticosteroids are allowed;
8. Known history of or seropositivity for Hepatitis B, Hepatitis C, or HIV;
9. Patients who have received live attenuated vaccines within 1 week of start of Everolimus and during the study. Patient should also avoid close contact with others who have received live attenuated vaccines. Examples of live attenuated vaccines include intranasal influenza, measles, mumps, rubella, oral polio, BCG, yellow fever, varicella and TY21a typhoid vaccines;
10. Patients who have a history of another primary malignancy, with the exceptions of:

    1. non-melanoma skin cancer,
    2. and carcinoma in situ of the cervix, uteri, or breast from which the patient has been disease free for ≥3 years;
11. Planned changes to concomitant medications;
12. Prior or concomitant therapy with known or possible anti-mTOR activity, including rapamycin (sirolimus);
13. Concomitant therapy with strong inhibitor (e.g., cyclosporine and ketoconazole) or inducer of CYP3A;
14. Active infection at time of enrollment;
15. Patients with a history of non-compliance to medical regimens or who are considered potentially unreliable or will not be able to complete the entire study;
16. Patients who are currently part of or have participated in any clinical investigation with an investigational drug within 1 month prior to dosing;
17. Pregnant or nursing (lactating) women;
18. Women of child-bearing potential (WOCBP), defined as all women physiologically capable of becoming pregnant, must use highly effective methods of contraception during the study and 8 weeks after. Highly effective contraception methods include:

    a. A combination of any two of the following: i. Use of oral, injected or implanted hormonal non-estrogen containing methods of contraception or; ii. Placement of an intrauterine device (IUD) or intrauterine system (IUS); iii. Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/ vaginal suppository; b. Total abstinence or; c. Male/female sterilization. Women are considered post-menopausal and not of child-bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks prior to randomization. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child-bearing potential.
19. Male patients whose sexual partner(s) are WOCBP who are not willing to use adequate contraception, during the study and for 8 weeks after the end of treatment
20. Major surgery, radiation therapy, or stereotactic radio-surgery within previous 4 weeks at time of screening
21. Neurosurgery within prior 6 months at time of screening.

Open-Label Inclusion Criteria

1. Patients who completed Double-Blind phase of the study and were assigned to the placebo treatment arm;
2. Verbal consent (and assent, as appropriate) obtained prior to any open-label phase study procedures.

Ages: 5 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2021-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Sahin, MD, PhD, Principal Investigator — Boston Children's Hospital
Locations (3):
- United States (3):
  - Stanford University, Palo Alto, California
  - Boston Children's Hospital, Boston, Massachusetts
  - Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with the National Database of Autism Research (NDAR)

REFERENCES:
- [Derived] Srivastava S, Jo B, Zhang B, Frazier T, Gallagher AS, Peck F, Levin AR, Mondal S, Li Z, Filip-Dhima R, Geisel G, Dies KA, Diplock A, Eng C, Hanna R, Sahin M, Hardan A; Developmental Synaptopathies Consortium. A randomized controlled trial of everolimus for neurocognitive symptoms in PTEN hamartoma tumor syndrome. Hum Mol Genet. 2022 Oct 10;31(20):3393-3404. doi: 10.1093/hmg/ddac111. PMID 35594551
- See also: Developmental Synaptopathies Consortium — http://www.rarediseasesnetwork.org/cms/dsc

RESULTS

PARTICIPANT FLOW:
Groups:
- RAD001: RAD001 is formulated as tablets of 5.0 mg or 2.5mg strength, blister-packed under aluminum foil in units of 10 tablets and dosed on a regular basis.
  RAD001: RAD001 is formulated as tablets of 5.0 mg strength, blister-packed under aluminum foil in units of 10 tablets and dosed on a regular basis. RAD001 tablets should be opened only at the time of administration as drug is both hygroscopic and light-sensitive.
  Patients will be instructed to take 4.5 mg/m2 of RAD001 orally with a glass of water at regular intervals at the same time in the morning after a light, nonfat breakfast.
- Placebo: Matching placebo will be provided as a matching tablet and will also be blister packed under aluminum foil in units of 10.
  Placebo: Matching placebo will be provided as a matching tablet and will also be blister packed under aluminum foil in units of 10. Matching placebo tablets should be opened only at the time of administration as drug is both hygroscopic and light-sensitive.
  Patients will be instructed to take 4.5 mg/m2 of the matching placebo orally with a glass of water at regular intervals at the same time in the morning after a light, nonfat breakfast.
Period: Overall Study
Arm/Group | RAD001 | Placebo
Started | 24 | 22
Completed | 21 | 20
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Investigator decision at baseline given safety concerns related to drug administration compliance | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RAD001 | Placebo | Total
Number analyzed (Participants) | 24 | 22 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.5 (11.3) | 14.7 (10.9) | 15.6 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 7 | 18
  Male | 13 | 15 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 20 | 18 | 38
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 2 | 2 | 4
Autism spectrum disorder (n) [Number; unit: participants] | 6 | 8 | 14
Autism spectrum disorder (%) [Number; unit: percentage of participants] | 25 | 36.3 | 30.4
Stanford-Binet Intelligence Scales, Fifth Edition (SB-5): Mean full scale IQ (FSIQ) [Mean (Standard Deviation); unit: scores on a scale] — FSIQ obtained from (SB-5) Stanford-Binet Intelligence Scales, Fifth Edition. FSIQ is a subscore of the SB-5. Scores range from 40-160, where a higher score number a better score (ie 40 is the worst, 160 is the best).
  scores on a scale | 77.8 (20.3) | 75.2 (23.5) | 76.6 (21.6)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability], Dropout
Description: The primary endpoint will be safety as measured by study drop-out rate due to side effects, comparing everolimus vs. placebo. We will also determine the frequency of adverse events by type and severity.
  This section displays participant dropout rate and for what reason.
Time Frame: Through study completion, an average of 6 months
Measure: Count of Participants; unit: Participants
Groups:
- RAD001: RAD001 is formulated as tablets of 5.0 mg or 2.5mg strength, blister-packed under aluminum foil in units of 10 tablets and dosed on a regular basis.
  RAD001: RAD001 is formulated as tablets of 5.0 mg strength, blister-packed under aluminum foil in units of 10 tablets and dosed on a regular basis. RAD001 tablets should be opened only at the time of administration as drug is both hygroscopic and light-sensitive.
  Patients will be instructed to take 4.5 mg/m2 of RAD001 orally with a glass of water at regular intervals at the same time (delete: each day) in the morning after a light, nonfat breakfast.
- Placebo: Matching placebo will be provided as a matching tablet and will also be blister packed under aluminum foil in units of 10.
  Placebo: Matching placebo will be provided as a matching tablet and will also be blister packed under aluminum foil in units of 10. Matching placebo tablets should be opened only at the time of administration as drug is both hygroscopic and light-sensitive.
  Patients will be instructed to take 4.5 mg/m2 of the matching placebo orally with a glass of water at regular intervals at the same time (delete: each day) in the morning after a light, nonfat breakfast.
- Total: Total Participants (RAD001 and Placebo groups)
Arm/Group | RAD001 | Placebo | Total
Number analyzed (Participants) | 24 | 22 | 46
Participants
  Dropout (Total) | 3 | 2 | 5
  Dropout due to participant/parent request | 2 | 1 | 3
  Dropout due to investigator request | 0 | 1 | 1
  Dropout due to other requests | 1 | 0 | 1

2. Primary Outcome: Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability], Adverse Events (AEs) Overview (% of Participants)
Description: The primary endpoint will be safety as measured by study drop-out rate due to side effects, comparing everolimus vs. placebo. We will also determine the frequency of adverse events by type and severity.
  this section displays the number of participants who experienced an AE and the description of such AEs, pertaining to:
  1. Seriousness
  2. Grade,
  3. Relation to treatment
  4. Recovery from AE
  5. Category
Time Frame: Through study completion, an average of 6 months
Measure: Number; unit: percentage of participants
Arm/Group | RAD001 | Placebo | Total
Number analyzed (Participants) | 24 | 22 | 46
percentage of participants
  Any AE (%) | 87.5 | 59.1 | 73.9
  Non-serious AEs (%) | 87.5 | 59.1 | 73.9
  Serious AEs (%) | 12.5 | 0 | 6.5
  Grade 1 (%) | 75 | 45.5 | 60.9
  Grade 2 (%) | 50 | 18.2 | 34.8
  Grade 3 (%) | 16.7 | 0 | 8.7
  Grade 4 (%) | 0 | 0 | 0
  Grade 5 (%) | 0 | 0 | 0
  Definitely not related to treatment (%) | 20.8 | 27.3 | 23.9
  Probably not related to treatment (%) | 37.5 | 18.2 | 28.3
  Possibly or probably related to treatment (%) | 70.8 | 31.8 | 52.2
  Definitely related to treatment (%) | 12.5 | 0 | 6.5
  Patients not recovered/not resolved from AEs (%) | 0 | 4.5 | 2.2
  Patients recovered/resolved with sequelae form AEs (%) | 4.2 | 0 | 2.2
  Patients recovered/resolved without sequelae fro AEs (%) | 83.3 | 59.1 | 71.7
  Patients recovering/resolving from AEs (%) | 8.3 | 3 | 4.3

3. Secondary Outcome: Change at 6 Months in Composite Score
Description: Composite score was based on the following:
  Stanford-Binet Intelligence Scales, 5th Ed (SB-5) non-verbal and verbal working memory standard score; for the SB-5, the minimum score is 40 and the maximum score is 160, where the higher score represents a better outcome.
  Conners' Continuous Performance Test, 3rd Ed (CPT-3) hit reaction time standard score (reverse coded; standard score generated from T-score); for the CPT-3, the min score is 0 and the max score is 90, where the lower the T-score, the better the outcome.
  Purdue Pegboard Test (PPT) both hands standard score (generated from T-score); for the PPT, the min score is 20 and the max score is 190, where the higher the T-score, the better the outcome.
  For the composite score, the higher the score, the better the outcome. The composite score is on the SS metric (M=100, SD=15, min=20, max=180).
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- RAD001 - Baseline; RAD001 - 6 Months: RAD001 is formulated as tablets of 5.0 mg or 2.5mg strength, blister-packed under aluminum foil in units of 10 tablets and dosed on a regular basis.
  RAD001: RAD001 is formulated as tablets of 5.0 mg strength, blister-packed under aluminum foil in units of 10 tablets and dosed on a regular basis. RAD001 tablets should be opened only at the time of administration as drug is both hygroscopic and light-sensitive.
  Patients will be instructed to take 4.5 mg/m2 of RAD001 orally with a glass of water at regular intervals at the same time in the morning after a light, nonfat breakfast.
- Placebo - Baseline; Placebo - 6 Months: Matching placebo will be provided as a matching tablet and will also be blister packed under aluminum foil in units of 10.
  Placebo: Matching placebo will be provided as a matching tablet and will also be blister packed under aluminum foil in units of 10. Matching placebo tablets should be opened only at the time of administration as drug is both hygroscopic and light-sensitive.
  Patients will be instructed to take 4.5 mg/m2 of the matching placebo orally with a glass of water at regular intervals at the same time in the morning after a light, nonfat breakfast.
Arm/Group | RAD001 - Baseline | Placebo - Baseline | RAD001 - 6 Months | Placebo - 6 Months
Number analyzed (Participants) | 24 | 22 | 21 | 20
score on a scale | 80.34 (15.23) | 75.14 (18.30) | 81.60 (17.17) | 78.47 (21.96)

4. Secondary Outcome: Change in Processing Speed at 6 Months, Conner's Continuous Performance Test (CPT)-3
Description: Processing speed will be evaluated using mean reaction time on the Conner's Continuous Performance Test (CPT)-3. This outcome evaluates the change from baseline to 6 months.
Time Frame: 6 months
Population: Change in processing speed scores were obtained from Conner's Continuous Performance Test (CPT)-3. Change in processing speed subscale scores were converted to standard scores, where a higher score indicates a better result (range 0-100).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAD001 - Baseline | Placebo - Baseline | RAD001 - 6 Months | Placebo - 6 Months
Number analyzed (Participants) | 24 | 22 | 21 | 20
score on a scale | 87.78 (20) | 86.30 (16.16) | 89.26 (22.35) | 90.15 (15.46)

5. Secondary Outcome: Change in Fine Motor Skills at 6 Months, Purdue Pegboard
Description: Fine motor skills will be evaluated using the Purdue Pegboard sub-tests average of both hands. This outcome evaluates the change from baseline to 6 months.
Time Frame: 6 months
Population: Change in fine motor skill scores were obtained from Purdue Pegboard. Fine motor skill scores were generated using standard scores, where a higher score indicates a better result (range 0-100).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAD001 - Baseline | Placebo - Baseline | RAD001 - 6 Months | Placebo - 6 Months
Number analyzed (Participants) | 24 | 22 | 21 | 20
score on a scale | 62.83 (20.52) | 55.92 (23.56) | 67.12 (20.08) | 61.49 (33.37)

6. Secondary Outcome: Change in Global Cognitive Ability at 6 Months, Stanford-Binet Intelligence Scales, Fifth Edition (SB-5) or Mullen Scales of Early Learning
Description: Change in global cognitive ability will be measured by Stanford-Binet 5 or Mullen; Full scale, verbal and nonverbal ability (IQ). This outcome evaluates the change from baseline to 6 months.
Time Frame: 6 months
Population: Global Cognitive Ability scores were obtained from Stanford Binet 5 or Mullen Scales of Early Learning depending on participant age and testing capability. Global Cognitive Ability subscale scores were converted to standard scores, where a higher score indicates a better result (range 0-100).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAD001 - Baseline | Placebo - Baseline | RAD001 - 6 Months | Placebo - 6 Months
Number analyzed (Participants) | 24 | 22 | 21 | 20
score on a scale
  Full Scale (FSIQ) | 77.83 (19.85) | 75.19 (22.90) | 79.39 (17.30) | 74.79 (25.79)
  Verbal (VIQ) | 78.79 (19.73) | 76.05 (23.67) | 78.46 (18.05) | 78.71 (27.07)
  Nonverbal (NVIQ) | 78.96 (19.03) | 75.91 (22.70) | 82.31 (16.25) | 73.15 (22.87)

7. Secondary Outcome: Change in Motor Functioning at 6 Months, Purdue Pegboard and Developmental Coordination Disorder Questionnaire (DCDQ)
Description: Motor functioning will be measured by the Purdue Pegboard (Pegs): Dominant and non-dominant hand combined standard scores and Developmental Coordination Disorder Questionnaire (DCDQ): Total score. This outcome evaluates the change from baseline to 6 months.
Time Frame: 6 months
Population: Change in motor functioning scores were obtained from Purdue Pegboard Developmental Coordination Disorder Questionnaire (DCDQ). Pegboard motor functioning scores were generated using standard scores, where a higher score indicates a better result (range 0-100). DCDQ motor functioning scores utilize the scale's total score, where higher scores indicate a better result (range 15-75).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAD001 - Baseline | Placebo - Baseline | RAD001 - 6 Months | Placebo - 6 Months
Number analyzed (Participants) | 24 | 22 | 21 | 20
score on a scale
  Purdue Pegboard (right hand) | 66.92 (22.83) | 58.64 (27.83) | 71.68 (30.18) | 61.47 (35.48)
  Purdue Pegboard (left hand) | 66.46 (23.02) | 61.82 (20.91) | 75.92 (24.76) | 60.26 (29.30)
  Purdue Pegboard (dominant hand) | 67.92 (21.92) | 58.63 (27.91) | 75.60 (24.78) | 59.25 (32.48)
  Purdue Pegboard (non-dominant hand) | 69.37 (21.92) | 61.89 (27.91) | 75.58 (24.78) | 62.36 (32.48)
  DCDQ Total Score | 37.51 (12.38) | 36.29 (14.20) | 40.01 (10.62) | 37.64 (16.37)

8. Secondary Outcome: Change in Memory, Executive Functioning, Autism Symptoms, Adaptive Behaviors, and Other Behaviors at 6 Months
Description: 1. Change in memory measured by Wide Range Assessment of Memory and Learning (WRAML-2) verbal learning core subtest, delayed recall, and recognition scaled scores over 6 months.
  2. Change in executive functioning measured by Behavior Rating Inventory of Executive Function (BRIEF-2) global executive composite standard score over 6 months.
  3. Change in autism symptoms measured by Social Responsiveness Scale (SRS-2) total standard score and Repetitive Behaviors Scale (RBS-R) total subscale score over 6 months.
  4. Change in adaptive behaviors measured by Vineland Adaptive Behavior Scales (VABS-III) adaptive behavior composite standard score over 6 months.
  5. Change in other behaviors measured by Child Behavior Checklist (CBCL) total problems standard score and Short Sensory Profile (SSP) total score over 6 months.
Time Frame: 6 months
Population: WRAML-2 scaled scores (range 1-19, higher = better) BRIEF-2 global executive composite standard score (range 0-100, higher = better) SRS-2 total standard score (range 0-100, higher = better) RBS-R total subscale score (range 0-56, LOWER = better) VABS-III adaptive behavior composite standard score (range 0-100, higher = better) CBCL total problems standard score (range 0-100, higher = better) SSP total score (range 38-190, higher = better)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAD001 - Baseline | Placebo - Baseline | RAD001 - 6 Months | Placebo - 6 Months
Number analyzed (Participants) | 24 | 22 | 21 | 20
score on a scale
  WRAML-2 verbal learning core subtest scaled score | 6.11 (2.65) | 6.90 (3.36) | 7.47 (3.93) | 7.22 (3.76)
  WRAML-2 verbal learning delayed recall scaled score | 6.73 (2.02) | 6.57 (3.40) | 8.13 (2.98) | 7.72 (2.99)
  WRAML-2 verbal learning recognition scaled score | 5.94 (3.49) | 5.97 (3.14) | 6.74 (3.96) | 6.42 (4.22)
  BRIEF-2 global executive composite standard score | 77.68 (19.77) | 71.18 (19.35) | 82.61 (17.43) | 74.24 (16.97)
  SRS-2 total standard score | 73.12 (18.23) | 67.52 (19.60) | 78.91 (17.75) | 66.90 (19.36)
  RBS-R total subscale score | 16.44 (16.83) | 23.35 (19.98) | 14.42 (5.86) | 19.96 (16.06)
  VABS-III adaptive behavior composite standard score | 76.96 (14.44) | 74.41 (18.21) | 81.56 (10.45) | 74.71 (15.75)
  CBCL total problems standard score | 85.90 (13.82) | 80.54 (18.07) | 90.10 (13.28) | 81.53 (14.80)
  SSP total score | 137.46 (21.68) | 128.25 (26.05) | 143.08 (16.54) | 126.52 (28.09)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | RAD001 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/22
Serious Adverse Events (participants affected / at risk) | 3/24 | 0/22
Other Adverse Events (participants affected / at risk) | 21/24 | 13/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RAD001 (N=24) | Placebo (N=22)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Renal lesions (Renal and urinary disorders) | 1 (1) | 0 (0)
Enterovirus infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RAD001 (N=24) | Placebo (N=22)
Stomatitis (General disorders) | 3 | 0
(Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Low Tolerance for Frustration (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Tremor (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 1
Middle Ear Inflammation (Ear and labyrinth disorders) | 2 | 0
External Ear Inflammation (Ear and labyrinth disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Runny Nose (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Stuffy Nose (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Mucositis Oral (Gastrointestinal disorders) | 7 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 1
Oral Pain (Gastrointestinal disorders) | 2 | 0
Oral Hemorrhage (Gastrointestinal disorders) | 1 | 0
Indigestion (Gastrointestinal disorders) | 0 | 1
Stomach Pain (Gastrointestinal disorders) | 1 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 1
Rash Acneiform (Skin and subcutaneous tissue disorders) | 2 | 0
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 2 | 0
Insect Bite (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Stomatitis (Skin and subcutaneous tissue disorders) | 4 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 1
Dry Skin Around Mouth (Skin and subcutaneous tissue disorders) | 0 | 1
Inflammatory Cystic Lesions (Skin and subcutaneous tissue disorders) | 1 | 0
Mouth Pain (Skin and subcutaneous tissue disorders) | 1 | 0
Bug Bite Induced Swelling (Skin and subcutaneous tissue disorders) | 1 | 0
Contact Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Cystic Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Bruising (Blood and lymphatic system disorders) | 1 | 0
Cholesterol, Triglycerides, HDL, And LD Out Of Range Clinically Significant (Blood and lymphatic system disorders) | 1 | 0
Easily Bruising (Blood and lymphatic system disorders) | 1 | 0
LDH Out Of Range Clinically Significant (Blood and lymphatic system disorders) | 1 | 0
Triglycerides And WBC Out Of Range Clinically Significant (Blood and lymphatic system disorders) | 1 | 0
Clinically Significant Out Of Range Labs (Blood and lymphatic system disorders) | 0 | 1
Gingival Bleeding (Blood and lymphatic system disorders) | 0 | 1
TSH, T4, And WBC Out Of Range, Clinically Significant (Blood and lymphatic system disorders) | 0 | 1
WBC, RBC, Hematocrit, And Absolute Neutrophil Out Of Range, Clinically Significant (Blood and lymphatic system disorders) | 0 | 1
Joint Range Of Motion Decreased (Musculoskeletal and connective tissue disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Upper Respiratory Infection (Infections and infestations) | 1 | 0
Influenza Type A (Infections and infestations) | 1 | 0
Viral Illness (Infections and infestations) | 1 | 0
Flu: Diarrhea, Cough, Running Nose (Infections and infestations) | 0 | 1
Otitis Media (Infections and infestations) | 1 | 0
Wrist Fracture (Injury, poisoning and procedural complications) | 1 | 0

LIMITATIONS AND CAVEATS:
1) Small sample size, as recruitment is difficult for rare neurogenetic disorders. 2) A subset of participants was unable to complete all assessments, largely due to the COVID-19 pandemic. Amidst COVID-19 pandemic, participants completed instruments remotely when possible. CPT-3 hit reaction time had a sample size n<10 at the month 6 timepoint, while the other measures had reasonable sample sizes. 3) Enrollment numbers were insufficient to power subgroup analysis, such as participants with ASD.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-13): https://cdn.clinicaltrials.gov/large-docs/07/NCT02991807/Prot_SAP_000.pdf